CLINICAL TRIAL: NCT00244803
Title: Redistribution and Metabolic Change in HIV Infection: Protocol 2 (FRAM Fat 2)
Brief Title: Redistribution of Fat and Metabolic Change in HIV Infection: Protocol 2 (FRAM Fat 2)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 03-07-02-01
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; FRAM 1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV Positive FRAM 1 Participant

SUMMARY:
The purpose of this study is to learn whether HIV-infected patients have blood abnormalities which could lead to heart attack or stroke, and to find out what factors may contribute to these abnormalities.

DETAILED DESCRIPTION:
This research is being done to learn whether HIV-infected patients have abnormalities in their blood vessels that could eventually lead to heart attack or stroke (atherosclerosis), in how fat is distributed in their body and in how their body handles fat and sugars. If there are abnormalities, this study will also try to find out what factors may contribute to those abnormalitites.

People who participated in FRAM 1 may join FRAM 2.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* previous FRAM 1 participant
* HIV positive

Exclusion Criteria:

* Artificial knee or hip replacement or Harrington rod
* Metal objects in the body.Pregnancy
* Breastfeeding or less than 3 months after breastfeeding
* Weight more than 300 pound
* On insulin, pancreatic enzymes, or thioridazine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men or women 18-65 years old, previous FRAM 1 participant, HIV positive
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cofrancesco Jr., M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, The Clinical Trials Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lake JE, Wohl D, Scherzer R, Grunfeld C, Tien PC, Sidney S, Currier JS. Regional fat deposition and cardiovascular risk in HIV infection: the FRAM study. AIDS Care. 2011 Aug;23(8):929-38. doi: 10.1080/09540121.2010.543885. Epub 2011 Jun 24. PMID 21767228